CLINICAL TRIAL: NCT02323243
Title: Clinical Interest of the Temporary Urethral Stent Allium " Bulbar Urethral Stent " in the Treatment of Detrusor Sphincter Dyssynergia
Acronym: ALLIUM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.861
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Detrusor Striated Sphincter Dyssynergia (DSSD)
Keywords: Detrusor striated sphincter dyssynergia; Temporary urethral stent
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allium BUS (Experimental): Temporary urethral stent
  Interventions: Device: Allium " Bulbar Urethral Stent " (BUS) system

INTERVENTIONS:
Device: Allium " Bulbar Urethral Stent " (BUS) system

SUMMARY:
Detrusor striated sphincter dyssynergia (DSSD) is defined as the persistence or increasing of the striated sphincter activity during voiding and characterizes the spinal cord injuries located under the protuberance. The standard treatment for DSSD is medical, either pharmacological or by clean intermittent self-catheterisation (CISC). Some patients are unable to perform CISC and require alternative surgical techniques such as external sphincterotomy which is invasive, irreversible and with no adjustment period for the patient.

Urethral stents have been developed as an alternative to surgical sphincterotomy. Temporary stents provide a non-definitive treatment, especially for evolutionary pathologies, for patients refusing a destructive surgery (psychosocial impact), or for patients having not defined yet their therapeutic preference. The Allium company has developed the " Bulbar Urethral Stent " (BUS) system, which advantages are the possibility to perform the procedure under local anesthesia and to remove more easily the stent, with similar performances compared to the other devices. In order to quantify the interest of the BUS system, the investigators propose to perform a prospective study aimed at describing its technical and clinical results in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged more than 18 years old
* Presenting detrusor striated sphincter dyssynergia in the opinion of the investigator, based on clinical data and proven urodynamically
* Detrusor striated sphincter dyssynergia with identified neurological origin
* With contraindication or failure of the conventional treatments
* Accepting the principle of the prosthetic incontinentation
* Having given his signed consent to participate in the study
* Affiliated with a social security scheme or assimilated.

Exclusion Criteria:

* Minor patient or protected adult according to the terms of the law
* Presenting contraindications to local regional anaesthesia
* Presenting contraindications or a previous failure to the treatment by prosthetic sphincterotomy
* Unable to hold a penile sheath.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who perceive their voiding condition improved or very improved | One month after the surgical intervention
  The perception of voiding condition by the patient will be measured with a 5-point Likert Scale. The patient will have to define the voiding condition compared to the initial (pre-procedure), as: very worse, worse, non-changed, improved, or very improved

SECONDARY OUTCOMES:
Number of stents correctly positioned | Immediately after the surgical intervention
Number of stent migrations | 1 month, 3 months, 6 months and 12 months after the surgical intervention
Number of stent removals performed without hemorrhage | 12 months after the surgical intervention
Number of complications, i.e. symptomatic urinary tract infections, encrustations, stenosis and hematuria, need for re-intervention and removals of the stent | Up to 12 months after the surgical intervention
Post-void residual volume measured by retrograde urinary urethrocystography | At inclusion and 1 month, 3 months, 6 months and 12 months after the surgical intervention
Maximum detrusor pressure and maximum urethral closure pressure, measured during the urodynamic testing | At inclusion, 1 month, 3 months, 6 months and 12 months after the surgical intervention
QUALIVEEN short form score (approved in French) | At inclusion and 1 month, 3 months, 6 months and 12 months after the surgical intervention
Number of patients requesting a change in the voiding method, i.e. premature removal of the stent | Up to 12 months following the surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie-Urologie - Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Background] Matillon X, Terrier JE, Arnouil N, Lalloue F, Pic G, Ruffion A. [Temporary urethral stents ALLIUM BUS "BULBAR URETHRAL STENT" for the treatment of detrusor sphincter dyssynergia]. Prog Urol. 2016 Sep;26(9):532-7. doi: 10.1016/j.purol.2016.07.005. Epub 2016 Aug 24. French. PMID 27567746